CLINICAL TRIAL: NCT04302987
Title: VITAMIN D INTERVENTION IN INFANTS: Effects of Early Vitamin D Exposure on Childhood Health at 6 Years - a Follow-up Study
Brief Title: Vitamin D Intervention in Infants - 6 Years Follow-up (VIDI2)
Acronym: VIDI2
Status: Completed | Type: Observational
Sponsor: University of Helsinki (Other)
Responsible Party: Principal Investigator, Sture Andersson, Professor Sture Andersson, University of Helsinki
Other Study IDs: Helsinki University
Record Dates: First submitted 2020-02-24; First posted 2020-03-10 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Bone Strength; Growth; Body Composition; Infection; Allergic Diseases; Dental Health
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples, saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Exposure to vitamin D intervention in early life may have permanent effects on physiology and metabolism. Bone growth and mineralization, development of immunity, body composition and brain structure and functioning may be affected. The importance of a long-term surveillance includes follow-up of both beneficial but also harmful effects of vitamin D.

Vitamin D intervention in infants (VIDI) study was conducted in 2013-2016. VIDI study was a large randomized trial that aimed to evaluate effects of two vitamin D supplemental doses of daily 10 ug and 30 ug from the age 2 weeks until 2 years on bone strength, infections, immunity, allergy, atopy and asthma, neurologic and cognitive development, and genetic regulation of mineral homeostasis. Current study is a 6 Years Follow-up (VIDI2) study of the original VIDI trial.

Our focuses of interest in the follow-up are: bone strength, growth pattern, body composition, and morbidity due to infections and allergic diseases, and the development of immunity. Further, in addition to more classical associates of vitamin D, our aim is to continue to follow-up children's neurocognitive development and mental health. We will also focus on the effect of vitamin D supplementation on occurrence of molar-incisor hypomineralization, dental caries, and oral immunity.

ELIGIBILITY:
Inclusion Criteria:

All who participated in the original VIDI study until last study visit at the age of 2 years.

Exclusion criteria:

None

Ages: 6 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: In the original VIDI study the eligible infants were born at term (37 weeks and 0 days' to 42 weeks and 0 days' gestation), with a birth weight within 2 SDs of the mean for gestational age. Infants excluded were those requiring intravenous glucose, antibiotics, nasal continuous positive airway pressure treatment for more than 1 day, phototherapy for more than 3 days, or nasogastric tube feeding for more than 1 day and infants with seizures.
Sampling Method: Non-Probability Sample
Enrollment: 415 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2022-05-27 (Actual)

PRIMARY OUTCOMES:
Areal bone mineral quantity | 6.5 years
  Bone mineral quantity in milligrams per millimeter is measured by peripheral quantitative computed tomography (pQCT).
Volumetric bone mineral density | 6.5 years
  Bone mineral density in milligrams per cubic centimeter is measured by pQCT.
Cross-sectional area of the bone | 6.5 years
  Cross-sectional area of the bone in square millimeters is measured by pQCT.
Bone mineral quantity | 6.5 years
  Bone mineral quantity in grams is measured by dual-energy X-ray absorptiometry (DXA).
Bone mineral density | 6.5 years
  Bone mineral density in grams per centimeter squared is measured by DXA.
Serum intact parathyroid hormone | 6.5 years
  Serum intact parathyroid hormone concentration is measured from blood samples with the blood gas analyzer ABL 90 FLEX or ABL 835 FLEX.
Plasma ionized calcium | 6.5 years
  Plasma ionized calcium concentration is measured from blood samples with the blood gas analyzer ABL 90 FLEX or ABL 835 FLEX.
Plasma alkaline phosphatase | 6.5 years
  Plasma alkaline phosphatase concentration is measured from blood samples with photometric methods.
Serum C-telopeptide of type I collagen | 6.5 years
  Serum C-telopeptide of type I collagen is measured with competitive polyclonal antibody assay.
Plasma fibroblast growth factor 23 | 6.5 years
  Plasma intact and C-terminal fibroblast growth factor 23 is determined with enzyme-linked immunosorbent assay.
Morbidity due to infectious diseases | 6.5 years
  Morbidity due to infectious diseases in frequencies and type are to be collected via questionnaires filled in by parents.
Morbidity due to allergic diseases | 6.5 years
  Morbidity due to allergic diseases and symptoms are to be collected via questionnaires filled in by parents.
Weight | 6.5 years
  Weight in kilograms is measured with a Seca 285 digital measuring station.
Height | 6.5 years
  .Height in centimeters is measured with a Seca 285 digital measuring station
Fat mass | 6.5 years
  Fat mass in kilograms based on ohms is measured by InBody bioelectrical impedance analysis.
Fat-free mass | 6.5 years
  Fat-free mass in kilograms based on ohms is measured with InBody.

SECONDARY OUTCOMES:
High sensitivity C-reactive protein | 6.5 years
  High sensitivity C-reactive protein is measured with enzyme immunoassay.
Plasma matrix metalloproteinase 8 | 6.5 years
  Plasma matrix metalloproteinase 8 is analysed with time-resolved immunofluorometric assay.
Gene variants | 6.5 years
  Gene variants associated with vitamin D metabolism and primary outcomes are performed using Sanger-sequencing, Taqman and genome-wide SNP-arrays.
Epigenetic changes | 6.5 years
  Epigenetic changes associated with vitamin D metabolism and primary outcomes are performed using methylation assays.
Cognitive abilities | 6.5 years
  Cognitive abilities are measured with Wechsler Intelligence Scale for Children-IV. Scales are scored according to the manual and standardized total scores vary between 10 and 159. Higher scores present better performance.
Executive functioning | 6.5 years
  Executive functions are measured with performance based test called NEPSY-II. Scales are scored according to the manual. Higher scores represent better performance.
Psychiatric disorders and symptoms | 6.5 years
  Psychiatric disorders and symptoms are measured with parent-rated questionnaire: the Child behavioral checklist. Scales are scored according to the manual. Maximum and minimum values very between subscales scales. Higher scores represent worse outcomes, i.e. more psychiatric symptoms.
Attention deficient and hyperactivity symptoms | 6.5 years
  Attention deficient and hyperactivity symptoms are measured with parent rated 'ADHD Rating Scale IV'-questionnaire. Scales are scored according to the published guidelines and higher scores reflect more problems.
Autism spectrum disorders and symptoms | 6.5 years
  Parent-rated Autism Spectrum Screening Questionnaire is used to measure Autism spectrum disorders and symptoms. Scales are scored according to the published guidelines and higher scores reflect more problems.
Sleep | 6.5 years
  Sleep is measured using a parent rated Sleep Disturbance Scale for Children. Questionnaire is scored according to publishers guidelines and the minimum and maximum scores vary. Higher scores in disturbance scales present worse outcome whereas a longer time at sleep represents a better outcome.
Temperament | 6.5 years
  Temperament is measured using parent rated questionnaire 'The Children's Behavior Questionnaire'. Questionnaire is scored according to manual and the minimum and maximum scores vary by temperament dimension. Higher scores do not as such mean better or worse outcome.
Prevalence of molar-incisor hypomineralization | 6.5 years
  Clinical evaluation by dentist of tooth enamel opacities, posteruptive enamel breakdown, atypical restorations, and/or extractions of molars according to the European Academy of Paediatric Dentistry criteria
Prevalence of caries | 6.5 years
  Clinical evaluation by dentist as decayed or filled tooth surfaces.
Salivary matrix metalloproteinase 8 level | 6.5 years
  Salivary matrix metalloproteinase 8 is analysed with salivary sample test.
SARS-CoV-2 virus antibodies | 6,.5 years
  SARS-CoV-2 virus antibodies are measured from blood samples
SARS-CoV-2 virus | 6.5 years
  SARS-CoV-2 virus PCR is analyzed from saliva

CONTACTS AND LOCATIONS:
Overall Officials: Sture Andersson, MD, Principal Investigator — Helsinki University Central Hospital
Locations (1):
- Children's Hospital, Helsinki, Finland

REFERENCES:
- [Derived] Seppala V, Sandboge S, Holmlund-Suila E, Hauta-Alus H, Lintula S, Kajantie E, Makitie O, Andersson S, Raikkonen K, Heinonen K. Early life vitamin D and neurocognitive abilities at age 6-8 years: a randomized clinical trial and observational analysis. Eur Child Adolesc Psychiatry. 2025 Oct 10. doi: 10.1007/s00787-025-02891-7. Online ahead of print. PMID 41071326
- [Derived] Sandboge S, Raikkonen K, Lahti-Pulkkinen M, Hauta-Alus H, Holmlund-Suila E, Girchenko P, Kajantie E, Makitie O, Andersson S, Heinonen K. Effect of Vitamin D3 Supplementation in the First 2 Years of Life on Psychiatric Symptoms at Ages 6 to 8 Years: A Randomized Clinical Trial. JAMA Netw Open. 2023 May 1;6(5):e2314319. doi: 10.1001/jamanetworkopen.2023.14319. PMID 37204794